CLINICAL TRIAL: NCT04185415
Title: A Participant-Blind, Investigator-Blind, Placebo-Controlled, Phase 1b Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of UCB0107 in Study Participants With Progressive Supranuclear Palsy (PSP)
Brief Title: A Study to Test the Safety and Tolerability of UCB0107 in Study Participants With Progressive Supranuclear Palsy (PSP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PSP003; 2019-002377-61 (EudraCT Number)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive Supranuclear Palsy; UCB0107; Phase 1 study; PSP
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bepranemab (Experimental): Subjects will be randomized to receive bepranemab.
  Interventions: Drug: bepranemab
- Placebo (Placebo Comparator): Subjects will be randomized to receive Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bepranemab — bepranemab will be administered in a predefined dosage.
  * Pharmaceutical Form: Solution for infusion
  * Route of Administration: Intravenous
  Other Names: UCB0107
  Arms: bepranemab
Drug: Placebo — * Pharmaceutical Form: Solution for infusion
  * Concentration: 0.9% w/v sodium chloride aqueous solution
  * Route of Administration: Intravenous
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the safety and tolerability of UCB0107 in study participants with Progressive Supranuclear Palsy (PSP).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥40 years of age at the time of signing the informed consent
* Participants meet the criteria for possible or probable Progressive Supranuclear Palsy (PSP) Richardson's Syndrome according the Movement Disorder Society (MDS)-PSP criteria
* Participant is able to walk at least 5 steps with minimal or no assistance (stabilization of one arm or use of cane/walker)
* Participant has reliable caregiver support during the whole study period or the participant is able to independently follow the study protocol
* Participant is stable on all treatments for at least 2 weeks prior to the Baseline Visit
* Participant has a body mass index (BMI) within the range 16.0 to 32.0 kg/m^2 (inclusive)
* Participants can be male or female
* Participant (and caregiver or legal representative, if applicable) is capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the Informed Consent form (ICF) and in this protocol. Informed consent must be obtained before initiating any study procedures

Exclusion Criteria:

* Ongoing, recurrent, severe headaches, including migraines
* Evidence of any clinically significant neurological disorder (including any clinically significant abnormalities on the screening magnetic resonance imaging) other than Progressive Supranuclear Palsy (PSP)
* Participant has a lifetime history of suicide attempt, or has suicidal ideation with at least some intent to act in the past 12 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Screening/Baseline" version of the Columbia-suicide severity rating scale (C-SSRS) at Screening
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator or medical monitor, contraindicates participation in the study
* The following liver enzyme test results:

  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) are >2.0x upper limit of normal (ULN)
  * Bilirubin >1.5x ULN (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35 %)
* The mean QT interval value (corrected by Fredericia's formula for the heart rate, QTcF) of the 3 Screening ECGs is >450 msec for male participants or >470 msec for female participants or QTcF is >480 msec in participants with bundle branch block
* Abnormalities in lumbar spine previously known or determined by a Screening lumbar x-ray (if conducted) that may jeopardize the execution of the lumbar puncture
* Participant was previously treated with tau-protein targeting drugs and/or tau-protein targeting antibodies or vaccines.
* Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to the first dose

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) from Baseline to the last Visit | From Baseline up to Week 68
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (13):
- Belgium (2):
  - Psp003 40122, Edegem
  - Psp003 40002, Leuven
- Germany (4):
  - Psp003 40277, Bochum
  - Psp003 40276, Düsseldorf
  - Psp003 40278, Essen
  - Psp003 40024, Hanover
- Spain (4):
  - Psp003 40159, Barcelona
  - Psp003 40267, Barcelona
  - Psp003 40100, Madrid
  - Psp003 40268, Madrid
- United Kingdom (3):
  - Psp003 40166, London
  - Psp003 40175, London
  - Psp003 40165, Southampton

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.